CLINICAL TRIAL: NCT04985825
Title: Phase 2 Study of Imgatuzumab in Patients With Advanced Cutaneous Squamous Cell Carcinoma (I-PACE)
Brief Title: Imgatuzumab in Patients With Advanced Cutaneous Squamous Cell Carcinoma
Acronym: I-PACE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Pega-One S.A.S. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Organization: Centessa Pharmaceuticals plc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO-001; 2021-003262-12 (EudraCT Number)
Record Dates: First submitted 2021-07-20; First posted 2021-08-02 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: Cutaneous Squamous Cell Carcinoma; Epidermal Growth Factor Receptor; Antibody-dependent Cellular Cytotoxicity; Carcinoma; Cancer
MeSH Terms: conditions — Carcinoma; Neoplasms | interventions — imgatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imgatuzumab monotherapy (Experimental)
  Interventions: Drug: Imgatuzumab

INTERVENTIONS:
Drug: Imgatuzumab — Imgatuzumab administered as an intravenous infusion on Day 1 and Day 8 of the first 21-day cycle, and on Day 1 of each subsequent 14-day cycle.

SUMMARY:
This study will evaluate the anti-tumor activity, safety, tolerability, immunogenicity, pharmacokinetics, and pharmacodynamics of imgatuzumab, a monoclonal antibody against epidermal growth factor receptor (EGFR) with enhanced antibody-dependent cellular cytotoxicity (ADCC) in patients with advanced cutaneous squamous cell carcinoma (CSCC). Quality of life of patients treated with imgatuzumab will also be assessed.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of CSCC
* CSCC of advanced stage
* Males or females at least 18 years of age at the time of consent
* Signed informed consent provided prior to any study procedures
* Ability to and willing to understand informed consent and comply with protocol requirements and procedures
* No more than two prior lines of systemic treatment for advanced disease
* Patients must have at least one lesion that is considered as measurable according to the Study Response Criteria
* Eastern Cooperative Oncology Group performance status 0 or 1
* Adequate function of bone marrow, liver, kidneys
* Availability of tumor tissue sample (either an archival specimen or a fresh biopsy material) at Screening

Key Exclusion Criteria:

* Prior systemic treatment for advanced disease with any anti-EGFR agent
* Active central nervous system metastasis
* Systemic anti-cancer therapy within five half-lives or two weeks, whichever is shorter, prior to first dose of the study drug
* Persistent toxicities from previous systemic anti-neoplastic treatments
* Wide-field radiotherapy within four weeks, or focal radiation for analgesic purpose or for lytic lesions at risk of fracture within two weeks prior to first dose of the study drug, or no recovery from side effects of such intervention
* Major surgery within four weeks prior to first dose of the study drug, or no recovery from side effects of such intervention
* Active infection requiring therapy
* Concomitant use of systemic steroids at dose of >10 mg of prednisone or its equivalent per day
* Known or suspected allergy/hypersensitivity to the study drug or any component of the study drug, other monoclonal antibodies, premedication medicines
* Concurrent participation in another investigational therapeutic clinical trial
* Pregnant or breast-feeding females
* Mental or medical conditions that prevent the patient from giving informed consent or participating in the trial
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or the study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for enrollment in this study

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) assessed by the Independent Central Review Committee (ICRC) according to the Study Response Criteria | Up to 24 months
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR) assessed by the ICRC according to the Study Response Criteria

SECONDARY OUTCOMES:
Disease Control Rate (DCR) assessed by the ICRC according to the Study Response Criteria | Up to 24 months
  Proportion of patients achieving CR, PR or Stable Disease (SD) assessed by the ICRC according to the Study Response Criteria
ORR assessed by the investigator according to the Study Response Criteria | Up to 24 months
  Proportion of patients achieving CR or PR assessed by the investigator according to the Study Response Criteria
DCR assessed by the investigator according to the Study Response Criteria | Up to 24 months
  Proportion of patients achieving CR, PR or SD assessed by the investigator according to the Study Response Criteria
Progression-free Survival (PFS) assessed by the ICRC | Up to 24 months
  Time from date of start of treatment to date of the first progression documented by the ICRC
Duration of Response (DoR) assessed by the ICRC | Up to 24 months
  Time from date of first assessment of response (CR or PR) to date of the first progression documented by the ICRC
Duration of Stable Disease (DoSD) assessed by the ICRC | Up to 24 months
  Time from date of first assessment of SD to date of the first progression documented by the ICRC
PFS assessed by the investigator | Up to 24 months
  Time from date of start of treatment to date of the first progression documented by the investigator
DoR assessed by the investigator | Up to 24 months
  Time from date of first assessment of response (CR or PR) to date of the first progression documented by the investigator
DoSD assessed by the investigator | Up to 24 months
  Time from date of first assessment of SD to date of the first progression documented by the investigator
ORR assessed by the ICRC according to the immune Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 24 months
  Proportion of patients achieving CR or PR assessed by the ICRC according to the iRECIST
ORR assessed by the investigator according to the iRECIST | Up to 24 months
  Proportion of patients achieving CR or PR assessed by the investigator according to the iRECIST
DCR assessed by the ICRC according to the iRECIST | Up to 24 months
  Proportion of patients achieving CR, PR or SD assessed by the ICRC according to the iRECIST
DCR assessed by the investigator according to the iRECIST | Up to 24 months
  Proportion of patients achieving CR, PR or SD assessed by the investigator according to the iRECIST
PFS assessed by the ICRC according to the iRECIST | Up to 24 months
  Time from date of start of treatment to date of the first iRECIST progression documented by the ICRC
PFS assessed by the investigator according to the iRECIST | Up to 24 months
  Time from date of start of treatment to date of the first iRECIST progression documented by the investigator
DoR assessed by the ICRC according to the iRECIST | Up to 24 months
  Time from date of first assessment of response (CR or PR) to date of the first iRECIST progression documented by the ICRC
DoR assessed by the investigator according to the iRECIST | Up to 24 months
  Time from date of first assessment of response (CR or PR) to date of the first iRECIST progression documented by the investigator
DoSD assessed by the ICRC according to the iRECIST | Up to 24 months
  Time from date of first assessment of SD to date of the first iRECIST progression documented by the ICRC
DoSD assessed by the investigator according to the iRECIST | Up to 24 months
  Time from date of first assessment of SD to date of the first iRECIST progression documented by the investigator
Incidence of Adverse Events | Up to 24 months
  Safety and tolerability profile assessed by Common Terminology Criteria for Adverse Events v5.0
Frequency of dose interruptions and reductions | Up to 24 months
  Safety and tolerability profile assessed by frequency of dose interruptions and reductions
Duration of dose interruptions and reductions | Up to 24 months
  Safety and tolerability profile assessed by duration of dose interruptions and reductions
Concentrations of imgatuzumab-reactive antibodies | Up to 24 months
  Immunogenicity profile characterized by concentrations of imgatuzumab-reactive antibodies
Maximum observed concentration (C[max]) | Up to 24 months
  Pharmacokinetic profile characterized by the maximum observed concentration (C[max]) of imgatuzumab
Area under the curve (AUC) | Up to 24 months
  Pharmacokinetic profile characterized by the area under the curve (AUC) of imgatuzumab
Terminal half-life (t[1/2]) | Up to 24 months
  Pharmacokinetic profile characterized by the terminal half-life (t[1/2]) of imgatuzumab
Time to maximum concentration (Tmax) | Up to 24 months
  Pharmacokinetic profile characterized by the time to maximum concentration (Tmax) of imgatuzumab
Change in scores of patient-reported outcomes | Up to 24 months
  Quality of life assessed by change in scores of patient-reported outcomes in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Scores are transformed linearly to a zero to 100 scale. A higher score on the functional scale and the global Health related Quality of Life indicates better functioning

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Heeger, MD, PhD, Study Director — PegaOne S.A.S.

IPD SHARING:
Plan to Share IPD: No